CLINICAL TRIAL: NCT06254547
Title: Do Leaderboards Improve Self-regulated Training in a Gamified Dermoscopy Training App? A Randomized, Controlled Trial.
Brief Title: Leaderboard Influence on Self-Regulated Training in a Gamified Dermoscopy Training App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Sigrid I. P. Kristensen, Bsc.med, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DL_Leaderboard_MS_01
Record Dates: First submitted 2024-01-26; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Melanoma (Skin); Skin Cancer
Keywords: Education; Skin Cancer; Gamification; Leaderboard; Diagnostic Accuracy; Self-regulated learning
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational messages and leaderboard (Experimental): This group will receive daily reminders/motivational messages. They will be able to view their personal score and will be ranked on a daily updated leaderboard.
  Interventions: Other: Daily updated ranking on leaderboard
- Only motivational messages (Experimental): This group will receive daily reminders/motivational messages. They will be able to view their personal score, but they will not be ranked on a leaderboard.
  Interventions: Other: Daily motivational message
- Control (No Intervention): This group will be able to view their personal score, but will not be ranked on a leaderboard or receive daily reminders/motivational messages.

INTERVENTIONS:
Other: Daily updated ranking on leaderboard — The intervention will last for seven days. Participants will on day two through seven receive a group daily message using an internet-based messaging service and view a daily updated leaderboard ranking.
  Leaderboards will demonstrate participant's ranking in their respective group, participant's (anonymized) name, cumulative point total, total case amount, and current level. Participant ranking will be based on the cumulative point total. All groups will have continual access to their personal score.
  Participants will not receive further training encouragement to train in the app or interact with the research group beyond this, aside from technological aid.
  Arms: Motivational messages and leaderboard
Other: Daily motivational message — The intervention will last for seven days. Participants will on day two through seven receive a group daily message using an internet-based messaging service encouraging training.
  Participants will not receive further training encouragement to train in the app or interact with the research group beyond this, aside from technological aid.
  Arms: Only motivational messages

SUMMARY:
This study aims to examine the isolated effect of leaderboards (scoreboards) and daily training motivation on dermatology skill acquisition and training engagement within a gamified dermoscopy training platform.

Research Questions:

What is the effect of leaderboards and/or daily motivation on diagnostic accuracy? What is the effect of leaderboards and/or daily motivation on self-regulated learning: time spent training and case amount? What is the effect of leaderboards and/or daily motivation on training distribution?

Method:

150 danish medical students will upon inclusion and end of trial answer a Multiple Choice Questionnaire (MCQ).

Participants will be asked to download the gamified training platform onto their mobile devices. Within the app participants can access quizzes on a library of 10,000+ skin lesions combined with written educational modules on histopathological skin diagnosis. Participants receive instant feedback on quiz answered. Points are awarded for correct answers and removed for incorrect answers.

Participants will be randomized to one of three groups; either receiving no communication from the principal investigator, receiving a daily motivational message, or receiving a once daily updated leaderboard ranking participant's scores.

The intervention will last for seven days, followed by a 14-day washout period.

DETAILED DESCRIPTION:
Subjects will be recruited through advertisements in online forums for medical students across all four Danish medical schools.

Upon recruitment, subjects will be included via an on-boarding online meeting. They will be introduced to the study and the training platform, and will, if they choose to participate, complete a consent form, a questionnaire of baseline information (age, gender, university semester, dermatological experience) and a 12-case validated diagnostic pre-test.

Participants will be randomized to study groups via sequential block randomization.

The intervention will last for seven days. Depending on group randomization, participants will on day two through seven either receive a group daily message using an internet-based messaging service (see appendix) and view a daily updated leaderboard ranking, only receive the group daily message, or receive neither.

Within the app, participants are able to train dermoscopy diagnosis through sessions of 10 cases. If participants correctly diagnose 8/10 cases, they will progress to the next session with new 10 cases of a higher difficulty, and so on. If participants do not reach a certain diagnostic accuracy, they will repeat their current level with 10 new cases until they are able to progress. There are a total of 6 session levels. Each case is assigned a difficulty level from one to four, calculated based on the percentage of times it has been answered correctly by previous users. In each session, participants are presented with 40% cases at their current level, 20% of an easier difficulty, 20% of a higher difficulty, and 20% cases of an unspecified difficulty.

Participants will be awarded 2 points multiplied by case difficulty for each correct answer. 2 points, multiplied by case difficulty, will be taken away if participants assign a benign diagnosis to a malignant case, and 1 point, multiplied by case difficulty, if a malignant diagnosis is assigned to a benign case. Participants will receive 0 points if a case is correctly classified as benign or malignant, but the precise histological diagnosis is incorrectly guessed (For example guessing melanoma on a basal cell carcinoma case, or nevus on a case of dermatofibroma). Participants will be able to view points earned following each training session, as well as a cumulative total.

After the seven-day interventional period, participants will start a 14-day washout period, in which participants can train freely, but no group will receive either daily messages or have access to the leaderboard. After the washout period, participants will be asked to complete a validated 12-case retention test, supervised by a member of the research group in a virtual meeting.

As this project is an educational study comprising medical students, it does not fulfill the criteria described in the Danish Scientific Ethical Committees Act § 2, and does not require approval by the The Regional Ethical Committee of the Copenhagen Capital Region of Denmark. A waiver has been obtained by The Regional Ethical Committee of the Copenhagen Capital Region of Denmark (case nr. F-23075872) The research group considers this project ethically responsible.

ELIGIBILITY:
Inclusion Criteria:

* Medical student at a Danish university

Exclusion Criteria:

* Have not completed a university-level course on histology
* Have completed or are currently enrolled in a clinical university course in dermatology
* Prior experience with the app Dermloop Learn or equivalent experience via. courses or by using other training platforms for skin diagnosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Time spent training | Three weeks
  The participant's time spent with the platform, measured by the platform
Amount of cases | Three weeks
  The number of cases participants assign a diagnosis to, measured by the platform
Change in diagnostic accuracy | Three weeks
  Measured as a percentage of correctly diagnoses skin lesions in validated multiple choice questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martin Frendø, MD, PhD, Study Director — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Herlev Hospital, Herlev, Denmark